CLINICAL TRIAL: NCT06862414
Title: Application and Validation of a Smartphone-based Deep Learning System for Oral Potentially Malignant Disorders (OPMD) and Oral Cancer Screening
Brief Title: Application and Validation of a Smartphone-based Deep Learning System for Oral Potentially Malignant Disorders and Oral Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202204032RIND
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Cancer Screening; Oral Cancer; Oral Potentially Malignant Disorders
Keywords: Deep learning systems; Artificial Intelligence
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: An open, three-arm, randomized controlled trial will be done in a medical center in Northern Taiwan between Jan 2025 to Dec 2025
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A (Experimental): Deep learning system
  Interventions: Device: Smartphone-based deep learning system
- B (Active Comparator): Board-certified dentist with deep learning system
  Interventions: Device: Smartphone-based deep learning system
- C (Active Comparator): non-certified health providers (general practitioners) with deep learning system
  Interventions: Device: Smartphone-based deep learning system

INTERVENTIONS:
Device: Smartphone-based deep learning system — The smartphone-based deep learning system was trained using a dataset of over 50,000 white-light macroscopic images collected between 2006 and 2013 to develop the YOLOv7 model. Lesions were categorized into three referral grades: benign (green), potentially malignant (yellow), and malignant (red).

SUMMARY:
The goal of this clinical trial is to learn if smartphone-based deep learning system works to accurately detect oral potentially malignant disorders and oral cancer in adults. It will also learn about if it is as effective as assessments conducted by dentists and non-certified health provider.

We expect that the deep learning system will have higher sensitivity in detecting oral potentially malignant disorders and oral cancer, where as the dentists and non-certified health providers will exhibit higher specificity in screening.

Participants will be grouped into three arms: deep learning system (arm A) or board-certified dentist with deep learning system (arm B) or non-certified health providers (general practitioners) with deep learning system (arm C).

Oral cancer risk factors, such as habits of smoking or having chewed betel nut or alcohol drinking, would be recorded by anonymous questionnaires.

DETAILED DESCRIPTION:
Background:

Oral cancer remains one of the leading causes of cancer-related deaths in Taiwan and worldwide. Artificial intelligence has the potential to improve oral cancer screening, enabling early detection by addressing healthcare access issues with high-quality solutions.

Objective:

To validate the smartphone-based deep learning system's accuracy in detecting oral potentially malignant disorders (OPMD) and oral cancer, while also demonstrating it is as effective as assessments conducted by dentists and non-certified health providers.

Methods:

Design, Setting and Participants: An open, three-arm, randomized controlled trial will be done in a medical center in Northern Taiwan between Jan 2025 to Dec 2025. The trial will include subjects aged 18 years or older who visit the cancer screening center for all kinds of screening. Oral cancer risk factors, such as habits of smoking or having chewed betel nut or alcohol drinking, would be recorded by anonymous questionnaires.

Interventions: Eligible subjects would be randomized in a 1:1:1 ratio using a computer-generated randomization algorithm to deep learning system (arm A) or board-certified dentist with deep learning system (arm B) or non-certified health providers (general practitioners) with deep learning system (arm C). The deep learning system in arm B and C would only be used for subsequent comparison and would not assist manual interpretation.

Main Outcomes and Measures: The primary outcome is the sensitivity and specificity for the three referral grades (benign (green), potentially malignant (yellow), and malignant (red)) by the deep learning system, dentists and non-certified health providers. The area under the curve (AUC) for each receiver operating characteristic (ROC) curve will also be calculated. The secondary outcome is subjects' feedback of comfortability during exam and the time needed for assessment.

Anticipated Results:

We hypothesize that deep learning systems will have higher sensitivity in detecting OPMD and oral cancer, whereas dentists and general practitioners will exhibit higher specificity in screening. The results could assist us in enhancing the oral cancer screening promotion process.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18) visiting cancer screening center

Exclusion Criteria:

* Unable to cooperate to fully open mouth/ navigate tongue
* Unable to cooperate for the assessment

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 954 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and accuracy | Within 6 months
  The primary outcome is the sensitivity and specificity for the three referral grades (green, yellow and red) by the deep learning system, dentists and non-certified health providers. The area under the curve (AUC) for each receiver operating characteristic (ROC) curve will also be calculated.

SECONDARY OUTCOMES:
Questionnaire | Within 6 months
  The secondary outcome is subjects' feedback of comfortability during exam evaluated by the visual analog scale (VAS) (a score out of 10). The time needed for screening will also be recorded for the assessment of efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yi Cheng, MD, MSc, DrPH, Study Chair — Department of Family Medicine, College of Medicine and Hospital, National Taiwan University
Locations (1):
- Department of Family Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hsu Y, Chou CY, Huang YC, Liu YC, Lin YL, Zhong ZP, Liao JK, Lee JC, Chen HY, Lee JJ, Chen SJ. Oral mucosal lesions triage via YOLOv7 models. J Formos Med Assoc. 2025 Jul;124(7):621-627. doi: 10.1016/j.jfma.2024.07.010. Epub 2024 Jul 12. PMID 39003230
- [Background] Tanriver G, Soluk Tekkesin M, Ergen O. Automated Detection and Classification of Oral Lesions Using Deep Learning to Detect Oral Potentially Malignant Disorders. Cancers (Basel). 2021 Jun 2;13(11):2766. doi: 10.3390/cancers13112766. PMID 34199471
- [Background] Hegde S, Ajila V, Zhu W, Zeng C. Artificial intelligence in early diagnosis and prevention of oral cancer. Asia Pac J Oncol Nurs. 2022 Aug 24;9(12):100133. doi: 10.1016/j.apjon.2022.100133. eCollection 2022 Dec. PMID 36389623
- [Background] Ng SW, Syamim Syed Mohd Sobri SN, Zain RB, Kallarakkal TG, Amtha R, Wiranata Wong FA, Rimal J, Durward C, Chea C, Jayasinghe RD, Vatanasapt P, Saleha Binti Ibrahim Tamin N, Cheng LC, Mazlipah Binti Ismail S, Tepirou C, Ariff Bin Abdul Rahman Z, Rajendran S, Kanapathy J, Liew CS, Cheong SC. Barriers to early detection and management of oral cancer in the Asia Pacific region. J Health Serv Res Policy. 2022 Apr;27(2):133-140. doi: 10.1177/13558196211053110. Epub 2022 Jan 22. PMID 35068209
- [Background] Khanagar SB, Naik S, Al Kheraif AA, Vishwanathaiah S, Maganur PC, Alhazmi Y, Mushtaq S, Sarode SC, Sarode GS, Zanza A, Testarelli L, Patil S. Application and Performance of Artificial Intelligence Technology in Oral Cancer Diagnosis and Prediction of Prognosis: A Systematic Review. Diagnostics (Basel). 2021 May 31;11(6):1004. doi: 10.3390/diagnostics11061004. PMID 34072804
- [Background] Gigliotti J, Madathil S, Makhoul N. Delays in oral cavity cancer. Int J Oral Maxillofac Surg. 2019 Sep;48(9):1131-1137. doi: 10.1016/j.ijom.2019.02.015. Epub 2019 Mar 13. PMID 30878273
- [Background] Peacock ZS, Pogrel MA, Schmidt BL. Exploring the reasons for delay in treatment of oral cancer. J Am Dent Assoc. 2008 Oct;139(10):1346-52. doi: 10.14219/jada.archive.2008.0046. PMID 18832270
- [Background] R VC, C R, Sridhar P, Ramachandra C, Kumar M. Barriers related to Oral Cancer Screening, Diagnosis and Treatment in Karnataka, India. Gulf J Oncolog. 2023 Sep;1(43):19-24. PMID 37732523
- [Background] Gonzalez-Moles MA, Aguilar-Ruiz M, Ramos-Garcia P. Challenges in the Early Diagnosis of Oral Cancer, Evidence Gaps and Strategies for Improvement: A Scoping Review of Systematic Reviews. Cancers (Basel). 2022 Oct 10;14(19):4967. doi: 10.3390/cancers14194967. PMID 36230890
- [Background] Warnakulasuriya S, Kujan O, Aguirre-Urizar JM, Bagan JV, Gonzalez-Moles MA, Kerr AR, Lodi G, Mello FW, Monteiro L, Ogden GR, Sloan P, Johnson NW. Oral potentially malignant disorders: A consensus report from an international seminar on nomenclature and classification, convened by the WHO Collaborating Centre for Oral Cancer. Oral Dis. 2021 Nov;27(8):1862-1880. doi: 10.1111/odi.13704. Epub 2020 Nov 26. PMID 33128420
- [Background] Stathopoulos P, Smith WP. Analysis of Survival Rates Following Primary Surgery of 178 Consecutive Patients with Oral Cancer in a Large District General Hospital. J Maxillofac Oral Surg. 2017 Jun;16(2):158-163. doi: 10.1007/s12663-016-0937-z. Epub 2016 Jul 8. PMID 28439154